CLINICAL TRIAL: NCT00470496
Title: A Phase I Study of Surgery Plus Intraoperative Photodynamic Therapy (PDT) in Patients With Resectable, Primary or Recurrent Head and Neck Cancer
Brief Title: Photodynamic Therapy Using HPPH in Treating Patients Undergoing Surgery for Primary or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 74606; NCI-2010-01941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 74606 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Thyroid Cancer; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage I Adenoid Cystic Carcinoma of the Oral Cavity; Stage I Basal Cell Carcinoma of the Lip; Stage I Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage I Follicular Thyroid Cancer; Stage I Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage I Lymphoepithelioma of the Nasopharynx; Stage I Lymphoepithelioma of the Oropharynx; Stage I Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage I Mucoepidermoid Carcinoma of the Oral Cavity; Stage I Papillary Thyroid Cancer; Stage I Salivary Gland Cancer; Stage I Squamous Cell Carcinoma of the Hypopharynx; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Adenoid Cystic Carcinoma of the Oral Cavity; Stage II Basal Cell Carcinoma of the Lip; Stage II Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage II Follicular Thyroid Cancer; Stage II Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage II Lymphoepithelioma of the Nasopharynx; Stage II Lymphoepithelioma of the Oropharynx; Stage II Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage II Mucoepidermoid Carcinoma of the Oral Cavity; Stage II Papillary Thyroid Cancer; Stage II Salivary Gland Cancer; Stage II Squamous Cell Carcinoma of the Hypopharynx; Stage II Squamous Cell Carcinoma of the Larynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage II Verrucous Carcinoma of the Larynx; Stage II Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Surgical Procedures, Operative; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (intraoperative PDT) (Experimental): Patients receive HPPH IV over 1 hour on day 1. Patients undergo surgery followed by laser light exposure to the entire tumor bed on day 2.
  Interventions: Drug: HPPH; Drug: photodynamic therapy; Procedure: conventional surgery

INTERVENTIONS:
Drug: HPPH — Given IV
  Other Names: Photochlor
Drug: photodynamic therapy — Undergo laser light exposure
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic
Procedure: conventional surgery — Undergo surgery
  Other Names: surgery, conventional

SUMMARY:
This phase I trial studies the side effects and best dose of photodynamic therapy using HPPH in treating patients who are undergoing surgery for primary or recurrent head and neck cancer. Photodynamic therapy (PDT) uses a drug, such as HPPH, that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. Giving photodynamic therapy after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identifying the maximum tolerated dose (MTD) of PDT among 4 investigated light dose levels (30, 50, 60 and 75) in combination with surgery in patients with recurrent or primary head and neck cancers.

SECONDARY OBJECTIVES:

I. To make initial observations of efficacy (i.e., tumor recurrence rate) of adjuvant PDT in these patients.

II. To determine the HPPH uptake and distribution (when feasible) in recurrent resected specimens.

III. Observe for wound complications.

OUTLINE: This is a dose-escalation study of laser light.

Patients receive HPPH intravenously (IV) over 1 hour on day 1. Patients undergo surgery followed by laser light exposure to the entire tumor bed on day 2.

After the completion of study treatment, patients are followed up at 1 and 3 months and then periodically thereafter at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable primary or recurrent head and neck squamous cell carcinomas (HNSCC) who are undergoing surgery to resect the cancer; (operable patients whose disease can be removed surgically with the expectation of clear margins, without compromising vital structures, i.e. respectability is individually determined by the surgeon and is based on anatomic extent of disease as well as technical ability of the operator)
* Female patients must not be pregnant (documented by human chorionic gonadotropin [HCG] test) and must be practicing a medically acceptable form of birth control, be sterile or post-menopausal
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must sign an informed consent according to Food and Drug Administration (FDA) guidelines acceptable to the Roswell Park Cancer Institute (RPCI) Institutional Review Board (IRB)
* No radiation therapy, chemotherapy or other biological therapy for at least 30 days prior to PDT

Exclusion Criteria:

* Patients with unresectable tumors
* Porphyria or hypersensitivity to porphyrin or porphyrin-like compounds
* White blood cell (WBC) < 4,000
* Platelet count < 100,000
* Prothrombin time 1.5 times above the upper normal limit
* Total serum bilirubin > 2.0 mg/d
* Serum creatinine > 2 mg%
* Alkaline phosphatase (hepatic) > 3 times the upper normal limit
* Serum glutamic oxaloacetic transaminase (SGOT) > 3 times the upper normal limit
* Patients on concurrent chemotherapy or radiation therapy will be excluded
* Patients who have received radiation therapy, chemotherapy or other biological therapy during the past 30 days
* Has not recovered from toxicity of prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-10-19 (Actual); Primary Completion 2011-10-28 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of photodynamic therapy in which 1 of 6 patients experience dose-limiting toxicity | 30 days

SECONDARY OUTCOMES:
Time to tumor progression or recurrence | From baseline until objective tumor progression, assessed up to 5 years
Uptake and distribution of HPPH in resected tumor tissue | Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Arshad, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Rigual NR, Shafirstein G, Frustino J, Seshadri M, Cooper M, Wilding G, Sullivan MA, Henderson B. Adjuvant intraoperative photodynamic therapy in head and neck cancer. JAMA Otolaryngol Head Neck Surg. 2013 Jul;139(7):706-11. doi: 10.1001/jamaoto.2013.3387. PMID 23868427